CLINICAL TRIAL: NCT06641895
Title: A Single-Arm, Open-Label, Single-Dose Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of BBM-D101 Injection in Patients with Duchenne Muscular Dystrophy
Brief Title: Evaluation of the Safety and Efficacy of BBM-D101 to Treat Patients with Duchenne Muscular Dystrophy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Mianyi Biopharmaceutical Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Jiwen Wang, study chair, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBM041-IIT1001
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-10

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: Adeno-Associated Virus; gene therapy; Duchenne muscular dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single dose intravenous injection of BBM-D101 (Experimental)
  Interventions: Genetic: BBM-D101

INTERVENTIONS:
Genetic: BBM-D101 — BBM-D101 is a recombinant adeno-associated virus vector-based gene therapy for DMD treatment. It is a suspension for single intravenous (IV) infusion.

SUMMARY:
The purpose of the study is to assess the safety, tolerability, and efficacy of BBM-D101 to treat patients with Duchenne Muscular Dystrophy.

DETAILED DESCRIPTION:
This is a single-arm, open-label study to evaluate the safety, tolerability, efficacy, pharmacokinetic, pharmacodynamic, and immune response of BBM-D101 within 52 weeks after a single intravenous infusion in DMD boys, as well as the long-term safety and efficacy of BBM-D101 for up to 5 years post infusion.

BBM-D101 is gene addition therapy based on engineered AAV delivery therapeutic protein gene cassette into muscle for treating DMD. Therapeutic protein could mediate the dystrophin-associated protein complex to prevent muscular dystrophy and to rescue the function of muscle.

ELIGIBILITY:
Inclusion Criteria:

1. The legal guardian of the subject fully understands the purpose, nature, methods, and possible risks of the study, and signs a written informed consent form;
2. The study includes ambulatory male subjects who are at least 4 years old and less than 8 years old (4 years old ≤ age < 8 years old) ;
3. Genetically confirmed diagnosis of DMD;
4. Have at least 1 of the following typical clinical signs or laboratory abnormalities of DMD: proximal muscle weakness, waddling gait, pseudo gastrocnemius hypertrophy, Gower's sign, pterygoid scapula;
5. Ability to cooperate with motor assessment testing, magnetic resonance imaging (MRI) and muscle biopsy according to the requirements of the study.

Exclusion Criteria:

1. Hepatitis B surface antigen (HBsAg) positive, hepatitis B virus deoxyribonucleic acid (HBV-DNA) ≥1000U/mL, hepatitis C virus ribonucleic acid (HCV-RNA) positive or human immunodeficiency virus (HIV) positive;
2. Receiving antiviral therapy for hepatitis B, hepatitis C, HIV, etc.;
3. Left ventricular ejection fraction (LVEF) <50% or ≥ class III cardiac function defined by New York Heart Association (NYHA);
4. With severe or persistent arrhythmias and congenital heart disease.
5. The subject's preventive treatment/cardiomyopathy treatment changes within 1 month before the start of the study treatment;
6. With underlying liver disease, such as previous diagnosis of portal hypertension, splenomegaly, hepatic encephalopathy, or hepatic fibrosis ≥ stage 3; or nodules, cysts found by B-ultrasound in the past, or elevated alpha-fetoprotein in laboratory tests during the screening period, etc., and these abnormalities are judged by the investigator to be clinically significant;

Ages: 4 Years to 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) events | 12 weeks
  To access the numbers of DLT events determined by the Safety Data Review Committee (SRC) in DLT observation period after BBM-D101 injection infusion.
The incidence of adverse events (AEs) and serious adverse events (SAEs) | 52 weeks
  To assess the safety of BBM-D101 Injection by AEs and SAEs.

SECONDARY OUTCOMES:
Changes from baseline in the North Star Ambulatory Assessment (NSAA) | 52 weeks
  To assess changes in NSAA from baseline within 12 weeks, 26 weeks, and 52 weeks after BBM-D101 injection infusion; The NSAA is a scale that rates performance of various motor abilities in ambulant children with Duchenne Muscular Dystrophy and is used to monitor disease progression and treatment effects. The NSAA total score is defined as the sum of all 17items, ranging from 0 (worst) to 34 (best).
Changes from baseline in the time to ascend 10-meter walk/run test (10MWR) without assistance | 52 weeks
  To assess changes in 10MWR from baseline within 12 weeks, 26 weeks, and 52 weeks after BBM-D101 injection infusion
Changes from baseline in the time to ascend time to rise (TTR) without assistance without assistance | 52 weeks
  To assess changes in TTR from baseline within 12 weeks, 26 weeks, and 52 weeks after BBM-D101 injection infusion
Changes from baseline in the time to ascend 4 steps (4-stair climb, 4SC) without assistance | 52 weeks
  To assess changes in 4-SC from baseline within 12 weeks, 26 weeks, and 52 weeks after BBM-D101 injection infusion
Changes from baseline in the time to ascend 100-meter walk/run test (100MWR) without assistance | 52 weeks
  To assess changes in 100MWR from baseline within 12 weeks, 26 weeks, and 52 weeks after BBM-D101 injection infusion
Changes from baseline in BBM-D101 genome copies in muscle biopsy samples | 52 weeks
  To assess changes of BBM-D101 genome from baseline in muscle in 12 weeks and 52 weeks following BBM-D101 administration. BBM-D101 genome was detected by Quantitative Polymerase Chain Reaction (QPCR).
Changes from baseline in BBM-D101 therapeutic protein level in muscle biopsy samples | 52 weeks
  To assess changes of BBM-D101 therapeutic protein from baseline in muscle in 12 weeks and 52 weeks following BBM-D101 administration. BBM-D101 therapeutic protein was detected by western blot (Jess) and tissue immunofluorescence.

CONTACTS AND LOCATIONS:
Overall Officials: Jiwen Wang, Study Chair — Shanghai Children's Medical Center, affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Children's Medical Center Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No